CLINICAL TRIAL: NCT06570837
Title: Iron Deficincy Among Children With type1 DM in Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Sayed Ahmed Sayed, Assistant Lecturer, Assiut University
Other Study IDs: Iron deficieny in type 1 DM
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Iron Deficiency, Anaemia in Children Type1DM
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Iron — observation effect of iron dificincy

SUMMARY:
detect the prevelance of anemic and non anemic iron deficiency in children with type 1 diabetes.assess the impact of anemic and non anemic iron deficiency in children with type 1 diabetes on their general condition

DETAILED DESCRIPTION:
Anemic and non anemic iron deficiency : is a global public health problem affecting both developing and developed countries with major consequences for human health as well as social and economic development.Iron deficiency anemia (IDA) appears to be more common in diabetic patients compared to non-diabetic population ,Iron deficiency (ID) and IDA can impair glucose homeostasis in human and may negatively affect glycemic control and predispose to more complications in diabetic patients. On the other hand diabetes and its complications are associated with anemia and its correction improves diabetes control and may prevent or delay the occurrence of complications. (1) Iron-deficiency anemia is the most common type of anemia. It occurs when your body doesn't have enough iron, which your body needs to make hemoglobin. When there isn't enough iron in your blood, the rest of your body can't get the amount of oxygen it needs.(2) Iron-deficiency anemia may be present without a person experiencing symptoms. (3) It tends to develop slowly; therefore the body has time to adapt, and the disease often goes unrecognized for some time. (4) If symptoms present, patients may present with the sign of pallor (reduced oxyhemoglobin in skin or mucous membranes),(5) and the symptoms of feeling tired, weak, dizziness, lightheadedness, poor physical exertion, headaches, decreased ability to concentrate, cold hands and feet, cold sensitivity, increased thirst and confusion. (6)(7) None of these symptoms (or any of the others below) are sensitive or specific. In severe cases, shortness of breath can occur. (8) Pica may also develop; of which consumption of ice, known as pagophagia, has been suggested to be the most specific for iron deficiency anemia.(9)

Iron deficiency without anaemia has been associated with:

* weakness, fatigue, reduced exercise performance, difficulty in concentrating, and poor work productivity(10)
* neurocognitive dysfunction including irritability(11)
* fibromyalgia syndrome(12)
* restless legs syndrome(13)
* symptom persistence in patients treated for hypothyroidism(14)
* poor neurodevelopmental outcomes in infants born to mothers with iron deficiency.(15)

Iron-deficiency anemia is confirmed by tests that include serum ferritin, serum iron level, serum transferrin, and total iron binding capacity. (16) A low serum ferritin is most commonly found. However, serum ferritin can be elevated by any type of chronic inflammation and thus is not consistently decreased in iron-deficiency anemia.(17) Serum iron levels may be measured, but serum iron concentration is not as reliable as the measurement of both serum iron and serum iron-binding protein levels. (18) The percentage of iron saturation (or transferrin saturation index or percent) can be measured by dividing the level of serum iron by total iron binding capacity and is a value that can help to confirm the diagnosis of iron-deficiency anemia; however, other conditions must also be considered, including other types of anemia.(19)

ELIGIBILITY:
Inclusion Criteria:

* Primary School age children with type 1 diabetes from 6 years up to 12year .

Exclusion Criteria:

- 1-All children with type1 diabetes less than 6 years and above 12 years. 2-Exclude other autoimmune diseases associated with diabetes mellitus (hypothyroidism, Addison disease , pernicious anemia, Celiac disease).

3-Any condition affecting iron metabolism.

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: cross sectional
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
detect the prevelance of anemic and non anemic iron deficiency in children with type 1 diabetes. | baseline
  detect the prevelance of anemic and non anemic iron deficiency in children with type 1 diabetes.

SECONDARY OUTCOMES:
assess the impact of anemic and non anemic iron deficiency in children with type 1 diabetes on their general condition | baseline
  assess the impact of anemic and non anemic iron deficiency in children with type 1 diabetes on their general condition

REFERENCES:
- [Background] Rubenstein MD, Wall RT. Clinical use of beta-thromboglobulin levels in diagnosing and treating consumptive and immune thrombocytopenia. Am J Hematol. 1981 Jun;10(4):369-73. doi: 10.1002/ajh.2830100406. PMID 6166192